CLINICAL TRIAL: NCT06433063
Title: Effect of 18F-Fluoromisonidazole (18F-FMISO) PET Imaging on Evaluation of Hypoxia Before Lu-177 PSMA Treatment for Prostate Cancer
Brief Title: Effect of Hypoxia on FMISO PET to Response to Lu-177 PSMA Treatment
Acronym: LuMISO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cigdem Soydal (Other)
Responsible Party: Sponsor-Investigator, Cigdem Soydal, Asc Prof of Nuclear Medicine, Ankara University
Organization: Ankara University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LuMISO
Record Dates: First submitted 2024-05-06; First posted 2024-05-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Prostatic Neoplasms; Hypoxia
MeSH Terms: conditions — Prostatic Neoplasms; Hypoxia

STUDY DESIGN:
Intervention Model Description: Metastatic castration resistant prostate cancer patients who will receive Lu-177 PSMA radionuclide treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment arm (Experimental): Patients who underwent FMISO PET imaging before Lu-177 PSMA radionuclide treatment for CRPC
  Interventions: Diagnostic Test: F-MISO PET

INTERVENTIONS:
Diagnostic Test: F-MISO PET — Evaluation of tumor hypoxia with F-MISO PET

SUMMARY:
It is aimed to evaluate hypoxia before Lu-177 PSMA treatment in prostate cancer and to show its effect on treatment success with 18F-FMISO PET imaging, which allows in-vivo evaluation and quantification of tumor hypoxia, which is known to be one of the factors affecting radiotherapy resistance.

DETAILED DESCRIPTION:
Prostate cancer is the second most common cancer in men and the fifth leading cause of cancer-related deaths. 20% of patients diagnosed with prostate cancer have metastatic disease, and survival rates of more than 5 years have been reported in only 26-30% of them. Androgen deprivation therapy (ADT) is the main treatment method used for years in the treatment of prostate cancer. However, a high rate of resistance develops to this treatment and becomes castration-resistant prostate cancer. Castration-resistant prostate cancer (CRPC) is defined as an increase in PSA levels, clinical or radiological progression, or the emergence of new distant metastases despite lowering serum testosterone to castration levels. FDA-approved drugs such as Sipuleucel-T, Docetaxel, Cabazitaxel, Abireterone, Enzalutamide, Radium-223, Rucaparib, and Olaparib have been shown to increase overall survival in mKDPK. Although there are many treatment classes that delay disease progression and increase survival, mKDPK remains incurable and fatal. Radionuclide therapy (Lu-177 PSMA) has emerged as a promising treatment in patients resistant to these treatments. Although some criteria have been defined to select patients who will benefit from treatment based on parameters such as SUVmax, some of the patients do not respond to radionuclide treatments, and PSA response can be achieved in only a little more than half of the patients in Lu-177 PSMA treatment, which stands out as one of the most effective therapies. The role of hypoxia, which is one of the possible factors affecting the treatment response other than PSMA avidity, in the success of Lu-177 PSMA treatment is currently unclear.

Radiation damage causing cell apoptosis and necrosis occurs through mechanisms such as ionizing radiation causing single or double chain breaks and creating reactive oxygen compounds in surrounding molecules. It is known that hypoxia causes radiotherapy resistance by preventing the formation of reactive oxygen compounds in tumors.

18F-Fluoromisonidazole (18F-FMISO) is an 18F-labelled PET radiopharmaceutical, like 18F-FDG, which has a half-life of 110 minutes and is frequently used in clinical practice. 18F-FMISO is a nitroimidazole class compound known to accumulate in hypoxic cells. After entering viable cells, 18F-FMISO is reduced to the RNO2 radical. In the presence of oxygen, 18F-FMISO can be oxidized again and freely exit the cell. However, since re-oxidation is not possible in hypoxic cells, 18F-FMISO is trapped in hypoxic but viable cells.

It has previously been shown that it is possible to predict radiotherapy response with 18F-FMISO PET imaging in malignancies such as head-neck and lung cancers and the feasibility of personalized treatment according to hypoxia demonstrated with 18F-FMISO. In a study, the presence of hypoxia was demonstrated with 18F-FMISO PET in high-grade tumors in patients receiving neoadjuvant ADT, and hypoxia was shown to regress with tumor response. However, to our knowledge, there is no study yet for Lu-177 PSMA treatment, which is one of the most important internal radiotherapies in prostate cancer. In this study, it was aimed to quantify hypoxia in primary tumors and metastases of prostate cancer with 18F-FMISO and to show its effect on treatment resistance.

Patients referred for Lu-177 PSMA treatment and found suitable for treatment will be included in the study. Within 4 weeks before Lu-177 PSMA treatment, patients will undergo PET imaging after 18F-FMISO injection and SUVmax, SUVmean, metabolic tumor volume and total 18F-FMISO retention parameters will be obtained from the tumors. Following this, patients will receive Lu-177 PSMA treatment in 4 cycles at 6-8 week intervals, as applied in standard clinical practice. Treatment response will be evaluated with Ga68 PSMA PET images taken after 4 cures of Lu-177 PSMA treatment. With 18F-FMISO findings, no changes will be made in the treatment process of the patients, and no additional imaging or examination will be performed after the treatment, other than routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years old
* Patients diagnosed with prostate cancer who were referred to our clinic for Lu-177 PSMA treatment and were found suitable for treatment

Exclusion Criteria:

* Has a life expectancy of less than 3 months
* ECOG>2
* contraindication for radionuclide treatment with Lu-177 PSMA

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate tumor hypoxia with F-MISO PET to PSA response | 6. month after radionuclide treatment
  Evaluation of the effect of tumor hypoxia to PSA response after Lu-177 PSMA treatment
To evaluate tumor hypoxia with F-MISO PET to radiological response | 6. month after radionuclide treatment
  Evaluation of the effect of tumor hypoxia to radiological response with RECIST criteria after Lu-177 PSMA treatment
To evaluate tumor hypoxia with F-MISO PET to PSMA PET response | 6. month after radionuclide treatment
  Evaluation of the effect of tumor hypoxia to PSMA response with RECIP criteria after Lu-177 PSMA treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University Medical School, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided